CLINICAL TRIAL: NCT06790186
Title: Improving Real-world Function for Persons with Schizophrenia (ImproFunc): a Single-case Experimental Design
Brief Title: Improving Real-world Function for Persons with Schizophrenia: a Single-case Experimental Design
Acronym: ImproFunc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 798582
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
Keywords: Cognitive difficulties
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Perceive, Recall, Plan and Perform (PRPP) intervention, to promote effective use of cognitive strategies for adults with schizophrenia when performing everyday activities in a real-world context. 27 persons with cognitive impairment due to schizophrenia will be included and provided the PRPP intervention in eight sessions. A single case experimental design with multiple baselines will be used to investigate the effectiveness of the PRPP intervention.
Masking Description: We plan for the assessor to be blinded when scoring the PRPP assessment. Therefore, one occupational therapist will conduct the assessments before and after the intervention, and another will provide the intervention for the participants. Additionally, to monitor observer drift , a third occupational therapist (the PhD candidate and the main supervisor) will be blinded to the phases and score 20 % of the PRPP assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perceive, Recall, Plan and Perform intervention (Other): Perceive, Recall, Plan and Perform (PRPP) intervention in promoting effective use of cognitive strategies for adults with schizophrenia in performing their daily activities will be given to all the included patients.
  Interventions: Behavioral: Perceive, Recall, Plan and Perform intervention Interventions:

INTERVENTIONS:
Behavioral: Perceive, Recall, Plan and Perform intervention Interventions: — The PRPP is a standardized system which determines the impact of information processing on performance of everyday activities. It is a method for assessment of performance mastery, and efficient use of cognitive strategies, as well as a model of intervention to train mastery and cognitive strategy use, in everyday activities. The PRPP assess task performance mastery, as well as cognitive strategy application

SUMMARY:
Existing treatment for individuals with psychosis primarily targets positive symptoms but has only modest effects on cognition and negative symptoms. Cognitive strategy training shows promising effects in reducing negative symptoms and increasing activity initiation in individuals with schizophrenia.

This project aims to investigate the effect of the Perceive, Recall, Plan and Perform (PRPP) intervention in promoting effective use of cognitive strategies for adults with schizophrenia in performing their daily activities. Twenty-seven individuals with schizophrenia will be recruited from Sykehuset Innlandet (Innlandet Hospital Trust) and assessed using PRPP prior to an eight-session PRPP intervention. Re-assessment will be conducted after the intervention, as well as at 3 and 6 months, to evaluate the long-term effects of the intervention. A single-case design will be used to investigate the intervention's effects. The primary outcome measure will be the PRPP assessment, and the secondary outcome measure will be the Goal Attainment Scale (GAS). Generalization measures will be used to evaluate whether there are relevant changes beyond the primary and secondary goals.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia, understand and speak Norwegian, live in their own community context, but are patients in Sykehuset Innlandet ( Innlandet Hospital Trust), either as outpatients or on discharge from inpatient care, a subjective experience of functional impairment and/or cognitive difficulties identified in an initial interview, and a stable state without any major medication change for at least two months before inclusion

Exclusion Criteria:

* Major physical disability, a current substance abuse problem, and cognitive deficits of organic origin or mental retardation

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
PRPP assessment | Assesments just after the intervention, as well as at 3 and 6 months
  Effective use of cognitive strategies in performing their daily activities

SECONDARY OUTCOMES:
Goal Attainment Scale | Assesments just after the intervention, as well as at 3 and 6 months
Health of the Nation Outcome Scale | Assesments just after the intervention, as well as at 3 and 6 months
Social Functioning Scale | Assesments just after the intervention, as well as at 3 and 6 months
Questionnaire about the Process of Recovery | Assesments just after the intervention, as well as at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Haug, PhD, Study Chair — Sykehuset Innlandet HF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin O. Rise of single-case experimental designs: A historical overview of the necessity of single-case methodology. Neuropsychol Rehabil. 2024 Apr;34(3):301-334. doi: 10.1080/09602011.2023.2181191. Epub 2023 Feb 22. PMID 36811612
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Aubin G, Stip E, Gelinas I, Rainville C, Chapparo C. Daily functioning and information-processing skills among persons with schizophrenia. Psychiatr Serv. 2009 Jun;60(6):817-22. doi: 10.1176/ps.2009.60.6.817. PMID 19487353
- [Background] Aubin G, Chapparo C, Gelinas I, Stip E, Rainville C. Use of the Perceive, Recall, Plan and Perform System of Task Analysis for persons with schizophrenia: a preliminary study. Aust Occup Ther J. 2009 Jun;56(3):189-99. doi: 10.1111/j.1440-1630.2007.00725.x. PMID 20854512
- [Background] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Effectiveness of the Perceive, Recall, Plan and Perform intervention for persons with brain injury in community-based rehabilitation: protocol for a single-case experimental design with multiple baselines. BMJ Open. 2022 Oct 5;12(10):e060206. doi: 10.1136/bmjopen-2021-060206. PMID 36198473
- [Background] Rocamora-Montenegro M, Compan-Gabucio LM, Garcia de la Hera M. Occupational therapy interventions for adults with severe mental illness: a scoping review. BMJ Open. 2021 Oct 29;11(10):e047467. doi: 10.1136/bmjopen-2020-047467. PMID 34716157
- [Background] Allott K, van-der-El K, Bryce S, Parrish EM, McGurk SR, Hetrick S, Bowie CR, Kidd S, Hamilton M, Killackey E, Velligan D. Compensatory Interventions for Cognitive Impairments in Psychosis: A Systematic Review and Meta-Analysis. Schizophr Bull. 2020 Jul 8;46(4):869-883. doi: 10.1093/schbul/sbz134. PMID 32052837
- [Background] Vita A, Barlati S, Ceraso A, Nibbio G, Ariu C, Deste G, Wykes T. Effectiveness, Core Elements, and Moderators of Response of Cognitive Remediation for Schizophrenia: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Psychiatry. 2021 Aug 1;78(8):848-858. doi: 10.1001/jamapsychiatry.2021.0620. PMID 33877289